CLINICAL TRIAL: NCT00308191
Title: A 6-Week Double-Blind, Parallel-Group, Active-Controlled Trial to Compare the Efficacy and Safety of Concomitant Treatment of Formoterol Fumarate Inhalation Solution 20 Mcg Twice Daily and Tiotropium 18 Mcg Once Daily to Tiotropium 18 Mcg Once Daily Alone in the Treatment of Patients With Chronic Obstructive Pulmonary Disease
Brief Title: A Phase IIIB Study to Compare the Efficacy and Safety of Concomitant Treatment in Patients With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dey (Industry)
Responsible Party: Director, Clinical Affairs, Dey L.P.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201-070
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2008-03

CONDITIONS: COPD
Keywords: COPD; Formoterol; Tiotropium
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate; Tiotropium Bromide

INTERVENTIONS:
Drug: Formoterol Fumarate
Drug: Tiotropium Bromide

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the concomitant treatment of formoterol fumarate with tiotropium bromide compared to treatment with tiotropium bromide alone.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of COPD
* Current or prior history of cigarette smoking

Exclusion Criteria:

* Medical diagnosis of asthma
* Significant condition or disease other than COPD

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128
Dates: Start 2006-04; Primary Completion 2006-05 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Measure of lung Function

SECONDARY OUTCOMES:
Change in lung function, vital signs; physical examinations; clinical laboratory assessments; adverse event reporting; patient questionnaires

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Research Site, Phoenix, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Sepulveda, California
  - Research Site, Walnut Creek, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Tamarac, Florida
  - Research Site, Gainesville, Georgia
  - Research Site, Auburn, Maine
  - Research Site, Ann Arbor, Michigan
  - Research Site, Livonia, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Liverpool, New York
  - Research Site, Rochester, New York
  - Research Site, Medford, Oregon
  - Research Site, Collegeville, Pennsylvania
  - Research Site, El Paso, Texas
  - Research Site, San Antonio, Texas

REFERENCES:
- [Result] Tashkin DP, Littner M, Andrews CP, Tomlinson L, Rinehart M, Denis-Mize K. Concomitant treatment with nebulized formoterol and tiotropium in subjects with COPD: a placebo-controlled trial. Respir Med. 2008 Apr;102(4):479-87. doi: 10.1016/j.rmed.2007.12.019. Epub 2008 Feb 6. PMID 18258423